CLINICAL TRIAL: NCT07270653
Title: Assessment of Tempromandibular Joint Changes After Treatment of Skeletal Class II Growing Patients by Twin Block Versus Monoblock
Brief Title: Assesment of Tempromandibular Joint ( TMJ ) Changes After Treatment of Skeletal Class II Cases by Twinblock vs Monoblock Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Fatema Mohamad, Principal investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORTO-108-2-G
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Skeletal Class II Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of skeletal class II by mandibular advancement using Twin block appliance (Experimental): Twinblock group
  Interventions: Device: twin block
- treatment of skeletal class II by mandibular advancement using Mono block appliance (Experimental): Monoblock group
  Interventions: Device: Mono block

INTERVENTIONS:
Device: twin block — Treatment of Skeletal class II by mandibular advancement using twinblock appliances ( removable myofunctional appliance)
  Arms: Treatment of skeletal class II by mandibular advancement using Twin block appliance
Device: Mono block — Treatment of Skeletal class II by mandibular advancement using Mono block appliances ( removable myofunctional appliance)
  Arms: treatment of skeletal class II by mandibular advancement using Mono block appliance

SUMMARY:
Assesment of TMJ changes after treatment of skeletal classII growing patients by Twinblock vs Mono block applinces

DETAILED DESCRIPTION:
Group (A): patients were treated by Twin block appliance Group (B): patients were treated by Mono block appliance

ELIGIBILITY:
Inclusion Criteria:

* skeletal class II malocclusion
* Defecient mandible
* ANB >4
* Growing female patients
* Age from 9-12 years

Exclusion Criteria:

* TMJ disease

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Tempromandibular changes including, condylar volume ( in cubic millimeters), length ( in millimeters) , height ( in millimeters) and position( in millimeters) | 8-12 months
  full skull CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Facility of dentistry, Alazhar university, girls branch, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Comparison of Skeletal Changes in the Temporomandibular Joint between the Twin Block Appliance and Fixed Functional Appliance: A Longitudinal Follow-up Study — https://pubmed.ncbi.nlm.nih.gov/38559857/